CLINICAL TRIAL: NCT01924572
Title: Placental Transfusion in Term Infants Placed Skin-to-Skin: A Pilot Controlled Trial
Brief Title: Placental Transfusion in Term Infants: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Judith S Mercer, Professor, Principal Investigator, University of Rhode Island
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Term Pilot Study
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Anemia
Keywords: umbilical cord clamping; Placental residual blood volume; hematocrit; hemoglobin; bilirubin
MeSH Terms: conditions — Anemia | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Immediate cord clamping (No Intervention): provider clamps and cuts the cord within 10 seconds after birth
- cord clamping at 2 minutes (Experimental): Provider places infant on maternal abdomen and cuts cord at 2 minutes after birth
  Interventions: Procedure: cord clamping at 2 minutes
- cord clamping at 5 minutes (Experimental): Provider places the infant on maternal abdomen and clamps and cuts cord at 5 minutes
  Interventions: Procedure: cord clamping at 5 minutes
- cord milking (Experimental): provider milks the cord 5 times from placenta to infant
  Interventions: Procedure: cord milking

INTERVENTIONS:
Procedure: cord clamping at 2 minutes
  Arms: cord clamping at 2 minutes
Procedure: cord clamping at 5 minutes
  Arms: cord clamping at 5 minutes
Procedure: cord milking
  Arms: cord milking

SUMMARY:
The proposed study is a pilot prospective controlled trial to measure the blood volume left in the placenta after varying cord clamping times when the infant is placed skin-to-skin on the maternal abdomen. Delaying cord clamping has been shown to decrease anemia in infants. However, the best way to get the most blood to the baby is not known. The practice of cord clamping at birth is not the same among doctors and midwives and we do not know the effect of putting he baby on the mother's abdomen.

DETAILED DESCRIPTION:
The proposed study is a pilot prospective controlled trial to measure the placental residual blood volume after varying cord clamping protocols when the infants are placed skin-to-skin on the maternal abdomen. The study assessed compliance of the providers with the different protocols. Placental transfusion (PT) has been shown to increase infant body iron stores at 6 months of age without increasing adverse outcomes. However, the optimal protocol to achieve adequate placental transfusion is not known. The practice of cord clamping at birth is not uniform among obstetrical providers because adequate evidence to support early or late cord clamping has been lacking.

Women were eligible to enroll in the study if they had no pregnancy complications, did not smoke, planned to breastfeed, and planned to deliver vaginally between 37 and 416/7 weeks. Women were enrolled prenatally on the labor and delivery unit. At birth, women were assigned to one of four cord clamping/milking groups. A cohort of infants with immediate cord clamping serves as reference group. Infants had blood samples drawn with the routine newborn screening blood samples done at 36 to 48 hours. Information on infant health and feeding was completed through an in-hospital visit to the mother and by home visit at two weeks of age. The primary outcome measures were placental residual blood volume and compliance with the various assigned cord clamping protocols. It was expected that infants with delayed cord clamping or cord milking would have less placental residual blood volume and that most providers would comply with the various random assignments.

ELIGIBILITY:
Inclusion Criteria: Women with normal pregnancy and presented at the labor room at 38-416/7 weeks for vaginal delivery; Intention to breast feed the babies; Consent for a follow up at 2 weeks of age

Exclusion Criteria: Abnormal pregnancy: Gestational or pre-existing diabetes, smoking and substance abuse, pre-eclampsia, fetal abnormality

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Placental Residual Blood volume | obtained immediately after birth
  Blood remaining in the placenta after cord clamping measured by drainage

SECONDARY OUTCOMES:
Infant hematocrit and hemoglobin | at 36 to 48 hours of age
  Capillary hematocrit and hemoglobin drawn when the genetic samples were drawn

OTHER OUTCOMES:
serum bilirubin | at 36 to 48 hours of age
  serum bilirubin drawn when the infant's genetic screen was drawn

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Mercer, PhD, CNM, Principal Investigator — University of Rhode Island; Debra A Erickson-owens, PhD, CNM, Study Director — University of Rhode Island
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States